CLINICAL TRIAL: NCT03699969
Title: A Clinical Study Comparing Hypofractionated Dose Escalated VMAT to Conventional CCRT in Locally Advanced Head and Neck Cancer
Brief Title: A Study Comparing Hypofractionated Dose Escalated VMAT to Conventional CCRT in Locally Advanced Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ehab Saad, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN12016
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Locally Advanced Head and Neck Cancer
Keywords: Hypofractionation; VMAT; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated dose escalated VMAT (Experimental): Hypofractionated dose escalated VMAT radiotherapy
  Interventions: Radiation: Hypofractionated dose escalated VMAT
- Conventional concurrent chemoradiation (No Intervention): Conventional concurrent chemoradiation

INTERVENTIONS:
Radiation: Hypofractionated dose escalated VMAT — measure the local control, progression free survival and overall survival
  Arms: Hypofractionated dose escalated VMAT

SUMMARY:
To compare efficacy and toxicity between hypofractionated dose escalated VMAT versus conventional concurrent chemoradiation in locally advanced head and neck cancer

DETAILED DESCRIPTION:
patients were randomized to receive either: 70Gy in 35fx in 7wks at 2Gy/fx concurrently with weekly cisplatin 40mg/m2 (Arm A) or 74Gy in 33 fractions (fx) in 6.5 weeks at 2.24Gy/fx (Arm B). Volumetric Modulated Arc Therapy (VMAT) plans were created for both treatment arms

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤70 years old.
2. Histopathologically confirmed squamous cell carcinoma of head and neck.
3. Locally advanced tumors (T3-T4 &/or N1-3) (stage IIB, III and stage IV-A: Staging by AJCC 7th edition).
4. Patients not exposed to radical surgery for current disease.
5. Performance status (ECOG) 2 or less.
6. No associated co-morbidity with contraindication to chemotherapy.
7. Normal Hemogram. (ANC ≥1.5x109/L, Platelets count ≥100x109/L, hemoglobin ≥80 g/L)
8. Accepted renal functions. (BUN & serum creatinine <1.5x upper limit of normal value with normal GFR).
9. Accepted liver functions. (total bilirubin and direct bilirubin < 1.5 x ULN & alanine aminotransferase and aspartate aminotransferase < 3 x ULN)
10. Informed consent.

Exclusion Criteria:

1. Patients with distant metastatic lesions, as detected by imaging techniques.
2. Patients with history of other head and neck malignancies.
3. Patients with history of previous head and neck irradiation.
4. Patients with a serious concomitant illness, such as active cardiac disease, severe uncontrolled hypertension, or uncontrolled infection.
5. Women who are pregnant or breast feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-15 (Estimated)

PRIMARY OUTCOMES:
Local control in the two arms | 33 months
  Local control by RECIST criteria

SECONDARY OUTCOMES:
The progression free survival in the two arms | 33 months
  The time (in months) from the end of radiotherapy to the date of first progression
The incidence of toxicity of radiotherapy by CTCAE protocol in the two arms | 33 months
  The number of patients who develop radiotherapy toxicity as assessed by CTCAE protocol Version 4.0

IPD SHARING:
Plan to Share IPD: No